CLINICAL TRIAL: NCT01448629
Title: An Open-labelled, Randomised, Controlled, Comparative, Explorative, Cross-over Study Investigating Safety and Performance of a New 1-piece Ostomy Product Compared Standard Care Ostomy Products in Subjects With Ileostomy
Brief Title: Safety and Performance of a New 1-piece Ostomy Product Compared to Standard Care Ostomy Products in Subjects Ileostomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn because of problems found with the baseplate
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP214OC
Record Dates: First submitted 2011-08-18; First posted 2011-10-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Leakage; Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- River (Experimental)
  Interventions: Device: River
- Standard Care (Active Comparator): Standard Care can have several manufacture and brand names. Standard Care is defined af the participants currently used stoma care product.
  Interventions: Device: Standard Care

INTERVENTIONS:
Device: Standard Care — Participants are using their own product and this procedure is called "Standard Care".
  Standard Care are the participants own products and may consist of several manufacturer and brand names.
  Arms: Standard Care
Device: River — River is a new developed product with Coloplast as manufacturer
  Arms: River

SUMMARY:
Introduction:

It is not an illness to have an ostomy, even though it is an indication of previous serious illness, such as cancer, which is the reason for approximately 80% of all ostomy operations. Ostomies can be divided into three categories: colostomy (large intestine), ileostomy (small intestine) and urostomy (urinary tract). All require surgical redirection of the intestine or urinary tract, allowing for elimination of urine and faeces by means of an opening in the abdominal wall. For the population included in this study, subject with an ileostomy, colitis ulcerosa is the main cause for an ileostomy where a surgical removal of the colon and rectum resulting in an ileostomy in theory cures the disease.

It can be very challenging to live with an ostomy and modern ostomy products should make life as easy as possible for people with ostomies.

Leakage and peristomal skin problems have been found to have a negative effect on the quality of life for people with ostomies. The skin problems are the reason for one out of three visits to ostomy nurses and occur much more frequently in people who have had ileostomies than in those who have had colostomies. It has been observed that the prevalence of peristomal skin problems is 21-60% among people who have ileostomies, 13-35% among those who have colostomies and 21-48% among those who have urostomies.

Leakage from ostomies that comes into contact with the skin is thought to predispose the patient to peristomal skin problems. One investigation of peristomal skin problems found that 77% of cases were related to contact with faeces or urine.

There are several reasons why leakage from an ostomy occurs, such as uneven peristomal area, improper handling of the ostomy product or a problematic ostomy (its formation, its location, retraction, prolapse or hernia). The ostomy may also change size with time, which can lead to leakage, if the ostomy products are not adapted accordingly. As a general rule, a check-up of the ostomy by an ostomy nurse or a doctor together with educational support can reduce these problems. Modern ostomy products should, however, also be constantly developed in order to lessen to the greatest extent possible the risk of leakage and associated inconveniences.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
List of Inclusion Criteria:

* Have given written informed consent.
* Are at least 18 years old.
* Have mental capacity to understand the study guidelines and questionnaires.
* Have had their ileostomy for at least 3 months
* Have an ileostomy with a diameter be-tween 19-40 mm.
* Are currently using a flat 1-piece product.
* Are able to change the product by them-selves or with help from a caregiver (e.g. spouse)
* Have experienced leakage under the base plate at least once a week over the last 2 weeks.

List of Exclusion criteria.

* Pregnant or breast-feeding.
* Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
* Currently using topical steroid product on peristomal skin (injections and oral treatment are accepted).
* Are currently using a convex product
* Participating in other clinical studies or have previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Leakage underneath the baseplate | two weeks

SECONDARY OUTCOMES:
Peristomal skin condition | Two weeks
  Measured by the Ostomy Skin Tool
Security | Two weeks
  The participants feeling of security when wearing the product, measured on a 5-point scale
Handling | Two weeks
  The participants ease of handling the products, measured on a 5-point scale
Comfort | Two weeks
  The participants feeling of comfort when wearing the product, measured on a 5-point scale
Adverse events | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol Katte, MD, Principal Investigator — Ashford and St. Peters Hospital